CLINICAL TRIAL: NCT06747520
Title: A Phase I Clinical Trial Assessing the Safety and Pharmacokinetics of a Single Intravenous Administration of Methoxetamine Hydrochloride in Subjects With Mild to Moderate Renal Impairment Compared to Individuals With Normal Renal Function
Brief Title: Phase 1 Renal Insufficiency Trial of Methoxyethyl Etomidate Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET-26-HCL-CP-004
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Renal Insufficiency
Keywords: Clinical Pharmacology; renal insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — ET-26 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild renal insufficiency（group A） (Experimental): 0.8mg/kg group
  Interventions: Drug: ET-26HCl
- moderate renal insufficiency（group B） (Experimental): 0.8mg/kg group
  Interventions: Drug: ET-26HCl
- normal renal function（group C） (Experimental): 0.8mg/kg group
  Interventions: Drug: ET-26HCl

INTERVENTIONS:
Drug: ET-26HCl — The dose is 0.8 mg/kg, single dose, Infusion time was 60s ± 5s.

SUMMARY:
Twenty-four subjects were divided into three groups: subjects with mild renal insufficiency, subjects with moderate renal insufficiency and subjects with normal renal function, with 8 subjects in each group.Subjects with mild renal insufficiency and moderate renal insufficiency were enrolled first, and then subjects with normal renal function were matched according to age, weight and gender. All patients received a single intravenous injection of 0.8mg/kg ET-26. To compare the pharmacokinetic characteristics of ET-26 and etomidate acid in subjects with mild and moderate renal insufficiency and normal renal function, and to provide clinical guidance for the use of ET-26 in patients with mild and moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

- All subjects

1. adult male and female subjects aged ≥18 years;
2. Body weight: body mass index (BMI) between 18.0 and 30.0 kg/m2 (including the cut-off value), with a body weight of at least 50 kg for male subjects and 45 kg for female subjects;
3. The subjects had good communication with the investigators, voluntarily signed the informed consent form and were able to complete the trial in accordance with the protocol; Subjects with renal insufficiency
4. The glomerular filtration rate (GFR) should meet the following criteria: mild renal insufficiency 60-89 mL/min (including both ends), moderate renal insufficiency subjects 30-59 mL/min (including both ends);
5. stable renal function with two absolute eGFR results (separated by at least 3 days) within the same CKD stage before administration;
6. no medication within 14 days before screening or with a stable medication regimen for renal impairment or other comorbidities (no adjustment in medication type, dose, or frequency for at least 2 weeks);
7. In addition to renal insufficiency and complications, the investigator judged the recipient's physical status according to medical history inquiry, physical examination, vital signs, cortisol test, laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function), and 12-lead electrocardiogram.

Subjects with normal renal function 8) matched with the renal insufficiency group by age (±10 years), weight (±15 kg), and gender (1:1); 9) GFR ≥90 mL/min; 10) normal or abnormal results of physical examination, vital signs, cortisol test, laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function), and 12-lead electrocardiogram without clinical significance.

Exclusion Criteria:

- All subjects

1. potentially difficult airway (modified Mallampati score III-IV);
2. hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody positive;
3. use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 14 days before screening;
4. a history of severe cardiovascular disease, including but not limited to organic heart disease, such as heart failure, myocardial infarction, angina pectoris, and malignant arrhythmia; Such as a history of torssion ventricular tachycardia, ventricular tachycardia, long QT syndrome or symptoms of long QT syndrome and family history (as indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes);
5. patients with severe infection, trauma, major surgery, or digestive system surgery within 1 month before screening that affect drug absorption;
6. those with allergic constitution, such as those with a known history of allergic to two or more substances; Or who, as judged by the investigator, may be allergic to the trial drug or its excipients;
7. binge drinking or regular drinking in the 6 months before screening, defined as drinking more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Or with a positive alcohol breath test at baseline;
8. smokers with an average of more than 5 cigarettes per day in the 3 months before screening or unable to quit smoking during the study;
9. those with drug abuse or drug use history within 3 months before screening; Or the baseline urine drug test was positive;
10. habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages and inability to quit during the trial;
11. those who have difficulty in blood collection or cannot tolerate blood collection by venipuncture;
12. participated in any other clinical trials (including drug and device clinical trials) within 3 months before screening;
13. vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
14. pregnant or lactating women;
15. those who plan to give birth or donate sperm during the trial and half a year after the completion of the trial, or those who do not agree that the subjects and their spouses should take strict contraceptive measures during the trial and half a year after the completion of the trial;
16. had blood loss or donation > 400 mL within 3 months before screening, or received blood transfusion within 1 month;
17. subjects with any factors considered by the investigator to be ineligible for the trial.

    Subjects with renal insufficiency
18. received a kidney transplant;
19. required renal dialysis during the study period;
20. urinary incontinence or anuria;
21. patients with acute disease of any organ other than the disease causing the diagnosis of renal insufficiency, and patients with any chronic disease (e.g., hepatic insufficiency) that could affect the internal course of the study drug were judged by the investigator to be ineligible for the trial;
22. abnormal coagulation function (INR>1.5 or prothrombin time (PT) >ULN+4 seconds or APTT>15×ULN), or clinically significant bleeding symptoms or clear bleeding tendency within 3 months before screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or receiving thrombolytic and anticoagulant therapy;
23. systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg at screening; The pulse was >100 bpm.

    Subjects with normal renal function
24. have a history of any clinically serious illness or disease or condition that the investigator considers may affect the trial results, including but not limited to a history of circulatory, respiratory, endocrine, nervous, digestive, urinary, or hematologic, immunologic, psychiatric, or metabolic diseases;
25. systolic blood pressure <90 mmHg or >139 mmHg, diastolic blood pressure <60 mmHg or >89 mmHg, and pulse <55 bpm or >100 bpm at screening;
26. have taken any prescribed medication within 14 days before dosing;
27. use of over-the-counter medicines, Chinese herbal medicines, or food supplements such as vitamins, calcium supplements within 7 days before administration;
28. cannot tolerate arterial blood sampling (e.g., Allen's test positive).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | up to 24 hours after infusion
  Cmax
Pharmacokinetic parameters | immediately after infusion to 24 hours after infusion
  AUC0-t
Pharmacokinetic parameters | up to 6 hours after infusion
  t1/2

SECONDARY OUTCOMES:
Pharmacodynamic indicators | MOAA/S score was measured three times within 60 minutes before administration as baseline value, was performed every 1 minute±5seconds for 5minutes after administration and every 2minutes±30seconds for 5minutes after administration
  Modified Observer"s Assessment of Alertness/Sedation（MOAA/S score）.The minimum score is 0 and the maximum is 5, with a score of 5 indicating that the subject is awake.The score was assessed multiple times throughout the procedure.
Pharmacodynamic indicators | BIS score was measured three times within 60 minutes before administration as baseline value,was performed every 1 minute±5seconds within 5minutes after administration, and every 2minutes±30seconds after 5minutes, until MOAA/S score ≥5
  Bispectral index(BIS score).The minimum score is 0 and the maximum is 100.The normal range of BIS scores is usually between 90 and 100, with higher values indicating greater brain activity and awareness.The score was assessed multiple times throughout the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Pharmaciae Doctor, Study Director — The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province), Jinan, Shandong, China